CLINICAL TRIAL: NCT06630000
Title: Focused Acceptance and Commitment Therapy (FACT) for Parents of Children With Pediatric Feeding Disorder
Brief Title: Focused Acceptance and Commitment Therapy (FACT)
Acronym: FACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dana Bakula, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00003127; K23MH133874 (NIH)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Feeding Disorders
Keywords: Feeding; Mental Health; Parents
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACT (Experimental): Behavioral: Focused Acceptance and Commitment Therapy (FACT) FACT is a 2-session intervention based on the Focused Acceptance and Commitment Therapy treatment literature
  Interventions: Behavioral: FACT
- Control (Active Comparator): The content of the control intervention covers a range of nutrition and healthy lifestyle topics including USDA's MyPlate
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: FACT — Two 90-minute FACT sessions led by a trained interventionist.
  Arms: FACT
Behavioral: Control — Two 90-minute sessions individually with a study interventionist, 2-weeks apart (focused on nutrition education).
  Arms: Control

SUMMARY:
This is a randomized clinical trial of Focused Acceptance and Commitment Therapy (FACT) vs. an attention-control condition (placebo) for improving the mental health of parents of children with pediatric feeding disorder.

The goal of this clinical trial is to compare two programs in parents of children with pediatric feeding disorders.

The main question[s] it aims to answer are:

FACT will result in clinically meaningful reductions in Mental Health(MH) problems among parents of children with Pediatric Feed Disorder (PFD) Identify factors that impact the feasibility of FACT delivery

Participants will asked to participate in one of two programs focused on parents of children with pediatric feeding disorders. The participants will also be asked to complete a battery of questionnaires at four timepoints during the study. The parents will be asked to video record a meal time three times during study.

Researchers will compare the FACT group with a control group to see if FACT will result in clinically meaningful change in parent stress and anxiety, and parent use of positive mealtime behaviors.

DETAILED DESCRIPTION:
The goal of this study is to advance the science of a brief parent mental health intervention for parents of children with pediatric feeding disorder using The goal of this study is to advance the science of a brief parent mental health intervention for parents of children with pediatric feeding disorder using The goal of this study is to advance the science of a brief parent mental health intervention for parents of children with pediatric feeding disorder using Focused Acceptance and Commitment Therapy (FACT) for Parents of Children with Pediatric Feeding Disorder. The ultimate goal of this research is to improve parent mental health and child health and feeding outcomes through a parent-focused behavioral intervention.

FACT is a 2-session acceptance and commitment therapy (ACT) intervention guided by Brown and Whittingham's ACT intervention for parents of children with neurodevelopmental conditions. Intervention content is based on principles of ACT, an evidence-based treatment for adult mental health problems. The intervention content is therefore broadly applicable to all parents but was specifically tailored for the needs of parents of children with neurodevelopmental conditions. In study phase 1 of this award, the investigators adapted parent ACT for parents of children with pediatric feeding disorder (PACT-F) with consultation from 2 parents of children with pediatric feeding disorder and 2 experts in parent ACT. The investigators now have a complete treatment package that has been tailored for parents of children with pediatric feeding disorder and is ready to be piloted.

This study will be conducted at a single site (Children's Mercy Hospital). The investigators will implement the clinical trial procedures and monitor feasibility success, and factors that may impact feasibility success. Participants who meet inclusion criteria will be randomized to either FACT or an attention control (control) condition. Participants will be blind to treatment condition (single blind study). The aim of the feasibility analyses is to evaluate factors critical to success, rather than evaluating whether the intervention is "feasible or not feasible". The aim of the proof-of-concept analyses is to determine if this intervention has promise and warrants a larger efficacy trial.

Parents randomized to FACT will complete two 90-minute FACT sessions individually with a study interventionist, 2 weeks apart. Parents randomized to the control group will complete two 90-minute sessions individually with a study interventionist, 2-weeks apart (focused on nutrition education). The control intervention will be parallel to the ACT intervention in all ways, including interactive components and the face-to-face time with health professionals (interventionists). The control condition intervention has already been developed by Dr. Davis's research team and covers a range of nutrition and healthy lifestyle topics including the United States Department of Agriculture's (USDA) MyPlate. An attention control condition was selected to mimic the interpersonal benefits that may come from meeting individually with a caring professional. The control condition intervention content (healthy lifestyles) was specifically chosen as it most closely reflects the types of information that parents would learn from healthcare professionals about the type of nutrition that their child needs. However, this type of intervention should not impact parent mental health.

Interventionists for both conditions will be individuals with at least master's degree training in mental health or a related field. The interventions will take via tele-video conferencing to allow participants to participate from home without needing transportation to and from the hospital. Both arms of the intervention will be manualized and interventionists in both arms will be trained using didactics and role playing with the Principle Investigator(PI). Intervention fidelity will be monitored by audio/video recording all sessions. The PI (Dr. Bakula) will review recordings each week and conduct separate 1-hour weekly supervision of study interventionists for each arm of the study (FACT & control).

Strategies will be used to promote fidelity in line with recommendations from the NIH Behavior Change Consortium. A fidelity checklist will be developed in line with adaptations to the intervention and will be piloted with study interventionists. The fidelity checklist will be refined during research team meetings. The fidelity checklist will be reviewed by the PI during supervision.

Hypothesis testing: The investigators will test the hypothesis that FACT results in clinically meaningful change using the Reliable Change Index (RCI; success defined as RCI > 1.96). The investigators anticipate that these procedures will be feasible, with feasibility success defined as recruitment rate above 60%, and retention, assessment completion, and intervention completion rate above 80%. Mixed methods data collection will identify factors that impact 1) recruitment rate (qualitative interviews, % meeting inclusion criteria, # of contact attempts), 2) retention rates (qualitative interviews, baseline characteristics; treatment group), 3) assessment completion rate (qualitative interviews, measure type), and 4) treatment completion rate (qualitative interviews, scheduling, treatment location).

ELIGIBILITY:
Inclusion Criteria:

* 1) Must be a parent aged 18+ (primary caregiver) of 2-6-year-old child with PFD
* 2) Child must be receiving outpatient PFD treatment at CMH
* 3) The parent must have a clinically significant elevation on at least one measure of parent MH (using established clinical cutoffs). Parents will be included regardless of whether the child has a new diagnosis or established diagnoses

Exclusion Criteria:

* 1) Parent has significant cognitive impairments
* 2) Parent does not speak English
* 3) Parent unable to obtain high speed internet at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | Baseline, 2 weeks post-intervention completion, 3-months post-intervention
  A 9-item self-report measure of depressive symptoms. Scores of 10 or more indicate probable depression.
General Anxiety Disorder (GAD-7) | Baseline, 2 weeks post-intervention completion, 3-months post-intervention
  A 7-item self-report measure of anxious symptoms. Scores of 10 or more indicate probable anxiety.
The Parent Psychological Flexibility Questionnaire (PPFQ) | Baseline, 2 weeks post-intervention completion, 3-months post-intervention
  19-item measure of psychological flexibility that is specific to parenting behaviors
Impact of Event Scale - Revised (IES-R) | Baseline, 2 weeks post-intervention completion, 3-months post-intervention
  A 22-item self-report measure of posttraumatic stress symptoms. Scores of 33 or more indicate clinically significant posttraumatic stress.
Perceived Stress Scale (PSS) | Baseline, 2 weeks post-intervention completion, 3-months post-intervention
  A 10-item self-report measure of perceived stress. Scores of 14 or more indicate clinically significant stress.
The Acceptance and Action Questionnaire (AAQ-2) | Baseline, 2 weeks post-intervention completion, 3-months post-intervention
  A 7-item self-report measure of psychological flexibility and experiential avoidance, which are targets of the behavioral treatment. Higher scores reflect more flexibility.
Behavioral Pediatrics Feeding Assessment Scale (BPFAS) | Baseline, 2 weeks post-intervention completion, 3-months post-intervention
  A 7-item self-report measure of psychological flexibility and experiential avoidance, which are targets of the behavioral treatment. Higher scores reflect higher probability of feeding disorder.
Early Childhood Parent Report Global Health 8a | Baseline, 2 weeks post-intervention completion, 3-months post-intervention
  An 8 item parent proxy measure of child overall health and skills. Scores of 40 or higher indicate moderate to severe symptoms/impairment.
Early Childhood Parent Report Self-Regulation - Flexibility 5a | Baseline, 2 weeks post-intervention completion, 3-months post-intervention
  A 5 item parent proxy measure of a child's ability to adapt to change. Lower scores indicate less ability to adapt to change.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No